CLINICAL TRIAL: NCT07292935
Title: Diagnostic Performance of Preoperative Gastric Ultrasound Compared to Gastroscopic Aspiration: A Prospective Clinical Study
Brief Title: Gastric Ultrasound Versus Gastroscopic Aspiration
Acronym: GUSGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Abdouli Hadhami, Docteur, Cheffe de clinique Adjointe en anesthésiologie, Hôpital Fribourgeois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GUSGA-2025
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Aspiration Risk; Full Stomach Status; Gastric Content
Keywords: Gastric Ultrasound; Gastroscopy; Estimated Gastric Volume; Preoperative Evaluation

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-group observational study in which all participants undergo both the index test (preoperative gastric ultrasound) and the reference standard (gastroscopy with complete aspiration). Gastric ultrasound is performed within one hour prior to gastroscopy. No randomization or parallel groups are involved. The study is designed to evaluate the diagnostic accuracy of ultrasound in detecting a full stomach and to compare estimated gastric volume with aspirated gastric volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric Ultrasound and Gastroscopy (Other): Single Group - Diagnostic Assessment
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — All enrolled participants undergo a preoperative gastric ultrasound within one hour prior to the scheduled gastroscopy. The gastric antrum is measured in standardized positions, and estimated gastric volume is calculated.

SUMMARY:
This is a prospective, single-center observational study conducted at the Fribourg Cantonal Hospital to evaluate the diagnostic performance of preoperative gastric ultrasound in determining gastric content and volume. Upper gastrointestinal endoscopy with complete suction of gastric contents serves as the reference standard.

Adult patients (≥ 18 years) scheduled for elective or urgent gastroscopy are consecutively recruited. A gastric ultrasound is performed within one hour before the endoscopic procedure. The antral cross-sectional area is measured in standardized positions (supine and right lateral decubitus), and gastric volume is estimated using validated formulas. Gastric content is categorized into three grades (empty, low-risk liquid content, or high-risk/solid content).

During gastroscopy, complete aspiration of gastric contents is performed at the start of the procedure. The aspirated volume and qualitative characteristics (liquid vs. solid) are recorded, and the stomach is classified as empty, partially full, or full by the endoscopist.

The primary objective is to determine the accuracy of gastric ultrasound in identifying a full stomach. Secondary objectives include evaluating the qualitative agreement between ultrasound and gastroscopy, correlating estimated gastric volume with aspirated volume, and identifying an optimal ultrasound-based volume threshold predictive of a full stomach.

Approximately 1,390 patients will be enrolled over one year to obtain at least 139 "full stomach" cases, based on prevalence estimates and sample size calculations. Statistical analyses will include diagnostic performance metrics, Cohen's kappa, correlation tests, Bland-Altman plots, and ROC curve analysis.

DETAILED DESCRIPTION:
Study Procedure and Conduct Each participant enrolled in the study will undergo a standardized two-step assessment protocol, consisting of a preoperative gastric ultrasound followed by a gastroscopy with complete aspiration of gastric contents. These procedures will be performed within a maximum interval of one hour, and conducted at Fribourg Cantonal Hospital within the Departments of Anesthesiology and Gastroenterology. All examinations will be performed by trained and credentialed operators, adhering to validated clinical protocols.

Following the acquisition of written informed consent, baseline demographic and clinical data will be collected. Gastric ultrasound will then be performed using a portable ultrasound device equipped with a low-frequency curvilinear transducer. The patient will be positioned sequentially in the supine and right lateral decubitus positions, with the upper body inclined at 45°, to obtain sagittal views of the gastric antrum. Antral diameters (antero-posterior and cranio-caudal) will be measured in each position, and the cross-sectional antral area (CSA) will be calculated accordingly. The estimated gastric volume (EGV) will be derived using the validated formula proposed by Perlas et al. Gastric contents will be classified into three qualitative grades (Grade 0 to 2), enabling stratification of aspiration risk.

Within one hour of the ultrasound, a diagnostic gastroscopy will be performed by an experienced gastroenterologist, following routine clinical practice. Immediately upon endoscope insertion and prior to any irrigation, complete aspiration of gastric contents will be performed to allow accurate measurement of the intragastric volume. The contents will be assessed macroscopically for appearance (e.g., clear, cloudy, bilious, alimentary) and consistency (liquid or solid). The aspirated volume will be quantified using a calibrated, graduated container. Based on visual assessment, the stomach will be classified as empty, partially full, or full.

All collected data will be documented using standardized case report forms and entered into a secure, anonymized database for subsequent statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* Indication for gastroscopy (scheduled or urgent), allowing complete aspiration of gastric contents
* Feasibility of performing gastric ultrasound within one hour prior to the endoscopic procedure
* Provision of written informed consent

Exclusion Criteria:

* Pregnancy
* History of major gastric or esophageal surgery
* Known disorders of gastric emptying (e.g., gastroparesis, gastric outlet obstruction)
* Cognitive impairment or language barriers preventing understanding of the study protocol
* Active vomiting or technical impossibility to aspirate gastric contents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1390 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
the diagnostic accuracy of gastric ultrasound in identifying a full stomach, using gastroscopy with aspiration as the reference standard. | Within 1 hour prior to gastroscopy
  Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and overall accuracy of preoperative gastric ultrasound in identifying a full stomach, compared to gastroscopy with complete aspiration of gastric contents. Gastric content is classified as empty, low-risk liquid content, or high-risk/solid content.

SECONDARY OUTCOMES:
Correlation coefficient between ultrasound-estimated gastric volume and aspirated gastric content volume during gastroscopy | Within 1 hour prior to gastroscopy
  Gastric volume is estimated by preoperative ultrasound and compared with the volume of gastric content aspirated during gastroscopy. The Pearson or Spearman correlation coefficient is calculated depending on data distribution.
Cohen's kappa coefficient for agreement between ultrasound and gastroscopy regarding gastric content nature | Within 1 hour prior to gastroscopy
  Agreement between gastric ultrasound and gastroscopy for classification of gastric content nature (clear liquid, turbid liquid, solid) is assessed using Cohen's kappa coefficient.
Optimal estimated gastric volume (EGV) threshold for predicting a full stomach | Within 1 hour prior to gastroscopy
  Determination of the optimal threshold of estimated gastric volume (EGV) measured by preoperative ultrasound for predicting a full stomach, using receiver operating characteristic (ROC) curve analysis. Sensitivity, specificity, and area under the ROC curve (AUC) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hadhami Abdouli, Docteur, Principal Investigator — Hôpital Cantonal Fribourgeois
Locations (1):
- HFR, Villars-sur-Glâne, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The shared individual participant data (IPD) will include only the data used in the publication of the study results, specifically:
  * Gastric ultrasound measurements (antral cross-sectional area, estimated gastric volume, gastric content grade)
  * Gastroscopy findings (aspirated gastric volume, qualitative gastric content classification)
  * Basic participant characteristics (age, sex, weight)
Supporting Information: Study Protocol, SAP
Time Frame: Starte Date: After publication of the study results End Date: 5 years after publication
Access Criteria: Researchers who submit a reasonable request for research purposes. Requests should be sent via email to the corresponding author. Access will be granted only after the request has been reviewed and approved by the study team.
  All shared data will be anonymized to protect participant confidentiality. The data and documents can be used solely for scientific research, and recipients are expected not to attempt to identify individual participants.